CLINICAL TRIAL: NCT04244578
Title: Transcranial Direct Current Stimulation in the Treatment of Dyslexia: a Randomized Double-blind Study.
Brief Title: Transcranial Direct Current Stimulation in the Treatment of Dyslexia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Deny Menghini, PhD, Clinical Psychologist, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 201201X002931
Record Dates: First submitted 2020-01-25; First posted 2020-01-28 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Dyslexia
Keywords: tDCS; transcranial direct current stimulation; transcranial electric stimulation; developmental dyslexia; specific learning disorders; treatment
MeSH Terms: conditions — Dyslexia; Specific Learning Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-Sham tDCS (Experimental): Each tDCS sessions will be delivered for 5 days for a total of non consecutive two weeks. The first session will be active tDCS and two months after, a sham tDCS will follow.
  Interventions: Device: Active tDCS; Device: Sham tDCS
- Sham-Active tDCS (Active Comparator): Each tDCS sessions (sham tDCS and active tDCS) will be delivered for 5 days for a total of non consecutive two weeks.
  The first session will be sham tDCS and two months after, an active tDCS will follow.
  Interventions: Device: Active tDCS; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active tDCS will be delivered to parieto-occipital areas for five consecutive days. tDCS will be delivered by a battery driven, direct current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands. The electrodes will be placed on the left (anodal) and right (cathodal) parieto-occipital areas, PO7 and PO8 position according to the 10-20 international EEG system for electrode placement. Stimulation intensity will be set at 1 milliampere (mA), the duration of stimulation will be 20 min.
  Other Names: Brainstim Active tDCS
Device: Sham tDCS — Sham tDCS will be delivered to parieto-occipital areas for five consecutive days. tDCS will be delivered by a battery driven, direct current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands. The electrodes will be placed on the left (anodal) and right (cathodal) parieto-occipital areas, PO7 and PO8 position according to the 10-20 international EEG system for electrode placement. Stimulation intensity will be set at 1 milliampere (mA), but the current will be applied for 30 s and will be ramped down without the participants awareness.
  Other Names: Brainstim Sham tDCS

SUMMARY:
The present study grounds on the absence of evidence-based treatment in individuals with dyslexia. At this topic, the present study will explore the potential effect of transcranial direct current stimulation (tDCS) over parieto-occipital brain regions, cerebral areas usually disrupted in individuals with dyslexia. tDCS will be administered without concomitantly training.

Therefore, the investigators hypothesized that active tDCS over parieto-occipital areas will enhance reading skills in children and adolescents with dyslexia. On the contrary, sham tDCS (placebo) over parieto-occipital areas will not have significant effect on reading. Further, both active and sham tDCS will be safe and well-tolerated.

DETAILED DESCRIPTION:
The study design is randomized stratified, cross-over, double-blind, placebo-controlled.

Children and adolescents with dyslexia will be selected and randomly assigned to two different groups: 1. Active tDCS over parieto-occipital areas + sham tDCS over parieto-occipital areas (Active-Sham tDCS); 2. Sham tDCS over parieto-occipital areas + active tDCS over parieto-occipital areas (Sham-Active tDCS).

In this project, the investigators will work to understand whether a brain-based intervention, with the use of tDCS without combined training, can enhance reading in individuals with dyslexia.

The protocol will allow the investigators to:

1. Testing the efficacy of stand-alone tDCS in enhancing reading in individuals with dyslexia;
2. Testing the critical role of brain regions (parieto-occipital areas) usually involved in reading and disrupted in dyslexia;
3. Predicting outcomes based on reading-related skills;
4. Investigating the safety and tolerability of tDCS;

The overarching goal is to provide a scientific foundation for devising new rehabilitation strategies in dyslexia.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with dyslexia (DSM-5, APA 2013)
* IQ ≥ 85

Exclusion Criteria:

* Having a comorbidity with an important medical conditions;
* Having neurological diseases;
* Having Epilepsy o family history of epilepsy;
* Receiving a treatment for dyslexia in the previous three months before the baseline screening;

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Non-word reading speed | up to one month after the end of the intervention
  The proportion of patients with change of at least 0.06 sill/sec in the non-word reading speed following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.

SECONDARY OUTCOMES:
Non-word reading accuracy | up to one month after the end of the intervention
  The proportion of patients with change in the non-word reading accuracy following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Word reading speed | up to one month after the end of the intervention
  The proportion of patients with change in the word reading speed following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Word reading accuracy | up to one month after the end of the intervention
  The proportion of patients with change in the word reading accuracy following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Text reading speed | up to one month after the end of the intervention
  The proportion of patients with change in the text reading speed following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Text reading accuracy | up to one month after the end of the intervention
  The proportion of patients with change in the text reading accuracy following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Verbal and visuo-spatial n-back | up to one month after the end of the intervention
  The proportion of patients with change in the index of verbal and visuo-spatial working memory (more score means better outcome) following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Phoneme Blending | up to one month after the end of the intervention
  The proportion of patients with change in the index of phoneme blending (more score means better outcome) following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Rapid Automatized Naming of color and letters | up to one month after the end of the intervention
  The proportion of patients with change in the accuracy and speed of Rapid Automatized Naming of color and letters following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Lexical Decision | up to one month after the end of the intervention
  The proportion of patients with change in the accuracy and speed of Lexical decision following Active tDCS sessions than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.
Questionnaire of safety and tolerability (Questionnaire of adverse effect) | up to one month after the end of the intervention
  The proportion of patients with change in the questionnaire of safety and tolerability (Questionnaire of adverse effect; Brunoni et al., 2011) following Active tDCS sessions will be the same than after Sham tDCS sessions both in ActiveSham tDCS and ShamActive tDCS.

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Hospital and Research Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Consensus Conference, Disturbi Specifici dell'apprendimento, ISS, 2011.
- [Background] Tressoldi P.E. L'evoluzione della lettura e scrittura dalla 2 elementare alla 3 media. Dati per un modello di sviluppo e per la diagnosi di disturbo specifico.Età Evolutiva, 53 - pp. 43-55, 1996
- [Background] Sartori G., Job R. e Tressoldi P.E. (2007), DDE-2. Batteria per la valutazione della dislessia e della disortografia evolutiva, Firenze, Organizzazioni Speciali.
- [Background] Cornoldi C. e Colpo G. (1998), Prove di Lettura MT per la Scuola Elementare-2, Firenze, Organizzazioni Speciali.
- [Background] Belacchi, C., Scalisi, T.G., Cannoni, E. e Cornoldi, C. (2008). Matrici Progressive di Raven Forma Colore (CPM-47). Manuale d'uso e standardizzazione italiana. Firenze, Organizzazioni Speciali.
- [Background] Achenbach, T.M., & Rescorla, L.A. (2001). Manual for the ASEBA School-Age Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Calvino, I. (1966). Marcovaldo ovvero le stagioni in città. Torino: Einaudi.
- [Result] Shaywitz BA, Shaywitz SE, Pugh KR, Mencl WE, Fulbright RK, Skudlarski P, Constable RT, Marchione KE, Fletcher JM, Lyon GR, Gore JC. Disruption of posterior brain systems for reading in children with developmental dyslexia. Biol Psychiatry. 2002 Jul 15;52(2):101-10. doi: 10.1016/s0006-3223(02)01365-3. PMID 12114001
- [Result] Temple E, Deutsch GK, Poldrack RA, Miller SL, Tallal P, Merzenich MM, Gabrieli JD. Neural deficits in children with dyslexia ameliorated by behavioral remediation: evidence from functional MRI. Proc Natl Acad Sci U S A. 2003 Mar 4;100(5):2860-5. doi: 10.1073/pnas.0030098100. Epub 2003 Feb 25. PMID 12604786
- [Result] Hoeft F, McCandliss BD, Black JM, Gantman A, Zakerani N, Hulme C, Lyytinen H, Whitfield-Gabrieli S, Glover GH, Reiss AL, Gabrieli JD. Neural systems predicting long-term outcome in dyslexia. Proc Natl Acad Sci U S A. 2011 Jan 4;108(1):361-6. doi: 10.1073/pnas.1008950108. Epub 2010 Dec 20. PMID 21173250
- [Result] Hoeft F, Hernandez A, McMillon G, Taylor-Hill H, Martindale JL, Meyler A, Keller TA, Siok WT, Deutsch GK, Just MA, Whitfield-Gabrieli S, Gabrieli JD. Neural basis of dyslexia: a comparison between dyslexic and nondyslexic children equated for reading ability. J Neurosci. 2006 Oct 18;26(42):10700-8. doi: 10.1523/JNEUROSCI.4931-05.2006. PMID 17050709
- [Result] Shaywitz SE, Shaywitz BA, Pugh KR, Fulbright RK, Constable RT, Mencl WE, Shankweiler DP, Liberman AM, Skudlarski P, Fletcher JM, Katz L, Marchione KE, Lacadie C, Gatenby C, Gore JC. Functional disruption in the organization of the brain for reading in dyslexia. Proc Natl Acad Sci U S A. 1998 Mar 3;95(5):2636-41. doi: 10.1073/pnas.95.5.2636. PMID 9482939
- [Result] Bakker DJ. Treatment of developmental dyslexia: a review. Pediatr Rehabil. 2006 Jan-Mar;9(1):3-13. doi: 10.1080/13638490500065392. PMID 16352500
- [Result] Simos PG, Fletcher JM, Bergman E, Breier JI, Foorman BR, Castillo EM, Davis RN, Fitzgerald M, Papanicolaou AC. Dyslexia-specific brain activation profile becomes normal following successful remedial training. Neurology. 2002 Apr 23;58(8):1203-13. doi: 10.1212/wnl.58.8.1203. PMID 11971088
- [Result] Stuss DT. The future of cognitive neurorehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):755-68. doi: 10.1080/09602011.2011.605590. Epub 2011 Sep 27. PMID 21950776
- [Result] Quintana H. Transcranial magnetic stimulation in persons younger than the age of 18. J ECT. 2005 Jun;21(2):88-95. doi: 10.1097/01.yct.0000162556.02720.58. PMID 15905749
- [Result] Jackson SR, Parkinson A, Manfredi V, Millon G, Hollis C, Jackson GM. Motor excitability is reduced prior to voluntary movements in children and adolescents with Tourette syndrome. J Neuropsychol. 2013 Mar;7(1):29-44. doi: 10.1111/j.1748-6653.2012.02033.x. Epub 2012 Jul 16. PMID 22804795
- [Result] Sokhadze EM, Baruth JM, Sears L, Sokhadze GE, El-Baz AS, Casanova MF. Prefrontal neuromodulation using rTMS improves error monitoring and correction function in autism. Appl Psychophysiol Biofeedback. 2012 Jun;37(2):91-102. doi: 10.1007/s10484-012-9182-5. PMID 22311204
- [Result] Croarkin PE, Wall CA, Lee J. Applications of transcranial magnetic stimulation (TMS) in child and adolescent psychiatry. Int Rev Psychiatry. 2011 Oct;23(5):445-53. doi: 10.3109/09540261.2011.623688. PMID 22200134
- [Result] Nitsche MA, Schauenburg A, Lang N, Liebetanz D, Exner C, Paulus W, Tergau F. Facilitation of implicit motor learning by weak transcranial direct current stimulation of the primary motor cortex in the human. J Cogn Neurosci. 2003 May 15;15(4):619-26. doi: 10.1162/089892903321662994. PMID 12803972
- [Result] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Result] Cattaneo Z, Pisoni A, Papagno C. Transcranial direct current stimulation over Broca's region improves phonemic and semantic fluency in healthy individuals. Neuroscience. 2011 Jun 2;183:64-70. doi: 10.1016/j.neuroscience.2011.03.058. Epub 2011 Apr 6. PMID 21477637
- [Result] Schlaug G, Renga V, Nair D. Transcranial direct current stimulation in stroke recovery. Arch Neurol. 2008 Dec;65(12):1571-6. doi: 10.1001/archneur.65.12.1571. PMID 19064743
- [Result] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Result] Monti A, Cogiamanian F, Marceglia S, Ferrucci R, Mameli F, Mrakic-Sposta S, Vergari M, Zago S, Priori A. Improved naming after transcranial direct current stimulation in aphasia. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):451-3. doi: 10.1136/jnnp.2007.135277. Epub 2007 Dec 20. PMID 18096677
- [Result] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Result] Schneider HD, Hopp JP. The use of the Bilingual Aphasia Test for assessment and transcranial direct current stimulation to modulate language acquisition in minimally verbal children with autism. Clin Linguist Phon. 2011 Jun;25(6-7):640-54. doi: 10.3109/02699206.2011.570852. Epub 2011 Jun 1. PMID 21631313
- [Result] Vines BW, Norton AC, Schlaug G. Non-invasive brain stimulation enhances the effects of melodic intonation therapy. Front Psychol. 2011 Sep 26;2:230. doi: 10.3389/fpsyg.2011.00230. eCollection 2011. PMID 21980313
- [Result] Miniussi C, Rossini PM. Transcranial magnetic stimulation in cognitive rehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):579-601. doi: 10.1080/09602011.2011.562689. Epub 2011 Jun 24. PMID 21462081
- [Result] Costanzo F, Menghini D, Caltagirone C, Oliveri M, Vicari S. How to improve reading skills in dyslexics: the effect of high frequency rTMS. Neuropsychologia. 2013 Dec;51(14):2953-9. doi: 10.1016/j.neuropsychologia.2013.10.018. Epub 2013 Oct 31. PMID 24184439
- [Result] Costanzo F, Menghini D, Caltagirone C, Oliveri M, Vicari S. High frequency rTMS over the left parietal lobule increases non-word reading accuracy. Neuropsychologia. 2012 Sep;50(11):2645-51. doi: 10.1016/j.neuropsychologia.2012.07.017. Epub 2012 Jul 20. PMID 22820638
- [Result] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Result] Lang N, Siebner HR, Ward NS, Lee L, Nitsche MA, Paulus W, Rothwell JC, Lemon RN, Frackowiak RS. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? Eur J Neurosci. 2005 Jul;22(2):495-504. doi: 10.1111/j.1460-9568.2005.04233.x. PMID 16045502
- [Result] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427
- [Result] Schlaug G, Marchina S, Norton A. From Singing to Speaking: Why Singing May Lead to Recovery of Expressive Language Function in Patients with Broca's Aphasia. Music Percept. 2008 Apr 1;25(4):315-323. doi: 10.1525/MP.2008.25.4.315. PMID 21197418
- [Result] Rubio-Morell B, Rotenberg A, Hernandez-Exposito S, Pascual-Leone A. [The use of noninvasive brain stimulation in childhood psychiatric disorders: new diagnostic and therapeutic opportunities and challenges]. Rev Neurol. 2011 Aug 16;53(4):209-25. Spanish. PMID 21780073
- [Result] Jancke L, Cheetham M, Baumgartner T. Virtual reality and the role of the prefrontal cortex in adults and children. Front Neurosci. 2009 May 1;3(1):52-9. doi: 10.3389/neuro.01.006.2009. eCollection 2009 May. PMID 19753097
- [Result] Holt RL, Mikati MA. Care for child development: basic science rationale and effects of interventions. Pediatr Neurol. 2011 Apr;44(4):239-53. doi: 10.1016/j.pediatrneurol.2010.11.009. PMID 21397164
- [Result] Mattai A, Miller R, Weisinger B, Greenstein D, Bakalar J, Tossell J, David C, Wassermann EM, Rapoport J, Gogtay N. Tolerability of transcranial direct current stimulation in childhood-onset schizophrenia. Brain Stimul. 2011 Oct;4(4):275-80. doi: 10.1016/j.brs.2011.01.001. Epub 2011 Feb 1. PMID 22032743
- [Result] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Result] Barca L, Burani C, Arduino LS. Word naming times and psycholinguistic norms for Italian nouns. Behav Res Methods Instrum Comput. 2002 Aug;34(3):424-34. doi: 10.3758/bf03195471. PMID 12395559